CLINICAL TRIAL: NCT02299726
Title: Early Aldosterone Blockade in Acute Heart Failure: An Exploratory Safety Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not funded
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Vanderbilt University (Other); Wayne State University (Other)
Responsible Party: Principal Investigator, Peter Pang, Associate Professor, Indiana University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R34HL118350-01A1
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Acute Heart Failure
Keywords: acute heart failure; MRA; emergency department
MeSH Terms: conditions — Emergencies | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental): spironolactone
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): matching placebo to active study drug
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Spironolactone
  Arms: Active
Other: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
Over one million hospitalizations for acute heart failure (AHF) occur over every year in the United States, resulting in high mortality, re-hospitalizations, and incurred financial costs; yet nearly every attempt over the last 10 years to improve outcomes with novel therapies have all failed. In this proposal, we will study whether a generic drug known as a mineralocorticoid receptor antagonist (more commonly known as an aldosterone blocker), proven to reduce morbidity and mortality for chronic heart failure patients, is safe and feasible to give to AHF patients in the emergency department and during hospitalization for a total of 3 days. The results of this study will provide necessary and sufficient data to design an efficacy study in a larger population to test whether early use of a high-dose of mineralocorticoid receptor antagonists will reduce post-discharge morbidity and mortality.

DETAILED DESCRIPTION:
This clinical trial pilot study - Early Aldosterone Blockade in Acute Heart Failure: An Exploratory Safety Study - will explore the safety of early mineralocorticoid receptor blockade with high-dose spironolactone (100mg/daily), an oral mineralocorticoid receptor antagonist, versus placebo (both in addition to standard therapy), in patients admitted with acute heart failure (AHF) for 3 days. Aim 1 will answer the critical question that early mineralocorticoid receptor (MR) antagonism in AHF patients is sufficiently safe to move forward with a definitive trial. Aim 2 will demonstrate feasibility of patient enrollment and compliance with treatment throughout the study to inform future study design and enrollment projections. This study will provide the necessary and sufficient data in order to plan a larger, simple, definitive trial to test the hypothesis that early aldosterone blockade in AHF patients will reduce mortality and 30-day readmissions.

The primary endpoint for the pilot study will be the difference in incidence of mean change of serum potassium of a specific amount from baseline to 120 hours from initial dose between placebo vs. spironolactone treated subjects.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female, age ≥ 21 years

  * Primary reason for admission is acute heart failure requiring IV loop diuretic therapy either in the emergency department (ED) or within 6 hours after direct hospital admission.
  * Enrolled within 12 hours of first dose of IV loop diuretic therapy
  * BNP > 300 pg/mL and/or NT-ProBNP > 1200 pg/mL by local laboratory
  * At least 1 of the following: Jugular Venous Distention, Peripheral edema, Radiographic evidence of pulmonary congestion
  * Ejection Fraction ≤ 40% within past 12 months by any method
  * Able to take oral medications
  * Able to provide written informed consent
  * Agrees to a minimum of 3 blood draws up to 72 hours from randomization

Exclusion Criteria:

* • Potassium ≥ 4.8mEq

  * eGFR (by sMDRD) < 45 ml/min/1.73 m2 or a worsening by 50% or more compared to any measurement in the last 6 months or planned ultrafiltration
  * History of or planned organ transplantation of any kind within the next 90 days
  * Invasive mechanical ventilatory support (non-invasive positive pressure ventilation is allowed)
  * Cardiogenic shock and/or treatment or planned treatment with inotropic or vasopressor medications (e.g. dobutamine, dopamine, milrinone, norepinephrine) or intra-aortic balloon pump
  * Refractory, end-stage HF defined as subjects who are appropriate candidates for specialized treatment strategies, such as transplant, ventricular assist devices, continuous intravenous inotropic therapy, or hospice care
  * Co-morbid condition with an expected survival <6 months or active cancer
  * History of stroke, cardiac surgery, or ACS currently or within past 60 days
  * Temperature ≥101.5 degrees F
  * Severe valvular or liver disease
  * On digoxin or history of MRA allergy or adverse drug reaction
  * Women who are currently pregnant or report a recent pregnancy (last 60 days) or plan on becoming pregnant during the next 4 months
  * Participation in another drug or device trial in which the last dose of drug was within the past 30 days or an investigational medical device has been implanted

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Change in Potassium from baseline through 5 days | 5 days